CLINICAL TRIAL: NCT05797480
Title: Dry Needling for Women With Provoked Vestibulodynia: A Feasibility and Acceptability Randomized Controlled Study
Brief Title: Dry Needling for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Principal investigator, professor and researcher, director of the research laboratory in urogynecology, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-4686
Record Dates: First submitted 2023-02-27; First posted 2023-04-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Provoked Vestibulodynia
Keywords: Dyspareunia; Vulvodynia
MeSH Terms: conditions — Dyspareunia; Vulvodynia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Baseline evaluation - Randomization to real dry needling or sham dry needling (6 sessions for 6 consecutive weeks) - post-treatment evaluation (2-week post-treatment)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Real Dry needling (Experimental): 1 dry needling treatment per week for 6 consecutive weeks
  Interventions: Other: Real Dry needling
- Sham: Non penetrating dry needling (Sham Comparator): 1 non penetrating dry needling per week for 6 consecutive weeks
  Interventions: Other: Non penetrating dry needling

INTERVENTIONS:
Other: Real Dry needling — Real dry needling will be applied to the pelvic floor, hip and lower back muscles.
  Other Names: Needling
  Arms: Experimental: Real Dry needling
Other: Non penetrating dry needling — Sham non penetrating dry needling (fixed needle in an introducer tube) will be applied to the pelvic floor, hip and lower back muscles.
  Other Names: Sham; Control
  Arms: Sham: Non penetrating dry needling

SUMMARY:
This is a randomized and controlled study investigating the feasibility and acceptability of a dry needling treatment for women suffering from provoked vestibulodynia. Following their enrollment in the study, participants will undergo a gynecological examination for confirmation of their diagnoses of provoked vestibulodynia. Women diagnosed with provoked vestibulodynia will be randomized into the dry needling group or the sham-needle group. The dry needling group will receive 6 sessions of real dry needling for 6 consecutive weeks. The sham group will receive 6 sessions of sham needling for 6 consecutive weeks, using a validated sham-needle. Outcomes measures will be assessed at baseline and at post-treatment and will include: feasibility and acceptability variables, pain intensity and quality, pain during palpation and pressure pain threshold, psychosexual variables, perceived improvement and satisfaction after the treatment as well as pelvic floor muscle stiffness and function.

DETAILED DESCRIPTION:
Up to 18% of reproductive-aged women experience chronic pain in the vulvar region during sexual intercourse. This chronic pain condition is called vulvodynia. The main subtype of this pain condition is provoked vestibulodynia (PVD), which is characterized by a sharp or burning pain at the vaginal opening when there is a pressure applied to the vulvar vestibule or attempting vaginal penetration. Women suffering from PVD suffer from sexual dysfunctions, psychological distress and worsened quality of life. The treatment options currently available are still quite limited and some women still experience pain despite undertaking all options available. We, therefore, proposed a randomized and controlled study to investigate the feasibility and acceptability of a dry needling treatment for women suffering from PVD. Women diagnosed with provoked vestibulodynia will be randomized into the dry needling group or the sham-needle group. Participants and evaluators will be blinded. The dry needling group will receive 6 sessions of real dry needling for 6 consecutive weeks. For the first three sessions, the dry needling/or sham techniques will be aimed at the muscles of the trunk, lower back, hips and SI joints. For the last 3 treatment sessions, the dry needling/or sham techniques will aimed at the pelvic floor muscles. The sham group will receive the same 6 sessions of sham needling for 6 consecutive weeks, using a validated sham-needle. Outcomes measures will be assessed at baseline and 2 weeks post-treatment and will include: feasibility (adherence to treatment, retention rates, adverse effects, recruitment rates and data on dry needling (needles, # of insertions, pain related) and acceptability variables. Secondary outcomes will include pain intensity during intercourse (numeric scale) and quality (McGill pain questionnaire), pain during palpation and pressure pain threshold (Pressure algometer), psychosexual variables (sexual distress and sexual function), change in pain catastrophizing, change in quality of life in domains associated with chronic pelvic pain (Pelvic Pain Impact questionnaire, severity of symptoms related to central sensitization), perceived improvement and satisfaction after the treatment as well as pelvic floor muscle stiffness (shearwave elastography and dynamometric speculum)and function (dynamometric speculum), blinding efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of provoked vestibulodynia according to a standardised gynaecologic exam
* Moderate to severe pain (≥ 5/10) in at least 90% of sexual intercourses or attempted sexual intercourse for at least 3 months

Exclusion Criteria:

* Other causes of vulvo-vaginal pain (e.g., spontaneous vulvovaginal pain not related to sexual intercourse/contact, dermatological condition, herpes, vulvo-vaginal atrophy)
* Post-menopausal state
* Actual or past pregnancy in the last year
* Urogynecological conditions (e.g., pelvic organs prolapse (POP) ≥ 3, urinary/vaginal infection active or in the last 3 months)
* Previous vulvar, vaginal or pelvic surgery (e.g., vestibulectomy, corrective pelvic organs prolapse surgery)
* Prior use of dry needling or acupuncture treatments
* Fear of needles or any contraindication to needling therapies
* Changes of medication that could influence pain perception (e.g., analgesic, antidepressant) in the last 3 months
* Other medical conditions that could interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment sessions | Through treatment completion (session 1 to 6; 6 weeks of treatment)
  a. To determine feasibility, the patients' adherence to treatment sessions will be recorded (present vs absent) as well as reasons for non-attendance.
Adherence to treatment protocol | Through treatment completion (session 1 to 6; 6 weeks of treatment)
  a. To determine feasibility by assessing adherence to treatment sessions.
Retention rate | Baseline to Post-treatment assessment (2-week post-treatment)
  a. To determine feasibility by assessing the percentage of participants completing the post-treatment assessment. Reason for dropouts will be compiled
Adverse effects | Through treatment completion (session 1 to 6; 6 weeks of treatment)
  a. Adverse effects observed and reported will be documented at each treatment session and at the post-treatment assessment.
Adverse effects | Post-treatment assessment (2-week post-treatment)
  a. Adverse effects observed and reported will be documented at each treatment session and at the post-treatment assessment.
Recruitment rate | Baseline
  a. To determine feasibility by assessing the percentage of participants included versus the participants screened. The barriers and reasons for refusing to participate as well as the reasons for exclusion will be documented
Intervention Acceptability Questionnaire | Baseline
  a. The Intervention Acceptability Questionnaire will be used to assess the participants' acceptability of the interventions. This questionnaire consists of 6 items measured on a VAS scale (Minimum value: 0; Maximum Value: 10). Each item is analyzed separately, with a greater score meaning higher acceptability of the intervention.
Intervention Acceptability Questionnaire | After treatment session 3 (week 3)
  a. The Intervention Acceptability Questionnaire will be used to assess the participants' acceptability of the interventions. This questionnaire consists of 6 items measured on a VAS scale (Minimum value: 0; Maximum Value: 10). Each item is analyzed separately, with a greater score meaning higher acceptability of the intervention.
Intervention Acceptability Questionnaire | Post-treatment assessment (2-week post-treatment)
  a. The Intervention Acceptability Questionnaire will be used to assess the participants' acceptability of the interventions. This questionnaire consists of 6 items measured on a VAS scale (Minimum value: 0; Maximum Value: 10). Each item is analyzed separately, with a greater score meaning higher acceptability of the intervention.

SECONDARY OUTCOMES:
Change in pain intensity during intercourse | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in pain intensity during intercourse (Numerical Rating Scale (NRS)). Ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever.
Change in pain quality | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes on the sensory, affective, and evaluative components of pain (McGill-Melzack Questionnaire). Ranging from 0 to 78, higher scores mean worst outcome (higher pain).
Change in pain catastrophizing | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes on pain catastrophizing (Pain catastrophizing scale (PCS)). Ranging from 0 to 52, higher scores mean worse outcome (higher pain catastrophizing).
Change in fear of pain | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in fear of pain (Pain anxiety Symptoms Scale (PASS-20). Ranging from 0 to 100, higher scores mean worse outcome (higher fear of pain).
Change in sexual function | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in sexual function (Female Sexual Function Index - FSFI). Ranging from 2 to 36, lower scores mean wort outcome (low sexual function).
Change in sexual distress | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in sexual distress (Female Sexual Distress Scale - FSDS). Ranging from 0 to 52, higher scores mean worse outcome (higher sexually related distress).
Change in quality of life in the domains associated with chronic pelvic pain | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in quality of life Pelvic Pain Impact Questionnaire (PPIQ). Ranging from 0 to 32, higher scores mean worse outcome (less quality of life associated with pelvic pain).
Severity of symptoms related with central sensitization | Baseline to Post-treatment assessement (2-week post-treatment)
  To explore changes in symptoms related to central sensitization (Central Sensitization Inventory). Ranging from 0 to 100, a higher scores indicates higher central sensitivity.
Satisfaction with treatment | Post-treatment assessment (2-week post-treatment)
  To determine acceptability by measuring the participants' satisfaction with the treatment on a Numeric Rating Scale (NRS) ranging from 0 (completely dissatisfied) to 10 (complete satisfied).
Patient's global impression of change | Post-treatment assessment (2-week post-treatment)
  To examine patient self-reported improvement (Patient's Global Impression of Change). Ranging from "very much worse" to "very much improved" on a 7-point scale.
Blinding effectiveness | Post-treatment assessment (2-week post-treatment)
  To assess the feasibility of maintaining blinding to group allocation for the participants. Evaluated by asking the question: ''What treatment do you think you have received? ''
Changes in pelvic floor muscle stiffness | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in pelvic floor muscle stiffness (Shearwave elastography)
Changes in pelvic floor muscle function | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in pelvic floor muscle function (Dynamometric speculum)
Changes in pain at palpation | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes at intravaginal palpation of the internal obturators and the levator ani muscles following a standardized procedure (Numerical Rating Scale). Ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever.
Changes in pressure pain threshold | Baseline to Post-treatment assessment (2-week post-treatment)
  To explore changes in pressure pain threshold if predetermined areas of the pelvis (Wagner algometer)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Morin, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Research Center of the Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No